CLINICAL TRIAL: NCT01297608
Title: A Double Blinded Study to Examine the Effect of Coated Suppositories on Fecal Incontinence in Patients With Spinal Cord Injury
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: RDD Pharma Ltd (Industry)
Responsible Party: Nir Barak, RDD Pharma
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RDD 106
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Fecal Incontinenece

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment (Experimental)
  Interventions: Drug: caoted suppository; Drug: coated suppository
- placebo (Placebo Comparator)
  Interventions: Drug: coated suppository

INTERVENTIONS:
Drug: caoted suppository — coated suppository with active drug
  Arms: treatment
Drug: coated suppository — coated suppository with placebo

SUMMARY:
This is a double blinded cross over study. Approximately 20 spinal cord injury patients will be participating in this 4 weeks study.The primary outcome is difference in fecal incontinence as recorded in diaries, between the treatment period and the treatment period.

ELIGIBILITY:
Inclusion Criteria:

Signed written informed consent; Male or female subjects 18 to 55 years of age; Spinal cord lesion/disease/injury at any level at least 3 months from injury. FISI (Fecal Incontinence Severity Index) > 8 units. The patient is able to understand the treatment and is willing to comply with the prescribed regimen

Exclusion Criteria:

* Known allergy to experimental drug..
* Porphiria.
* Glaucoma.
* Pregnancy or lactation.
* Active or past history of cardiovascular or cerebrovascular disease including unstable angina, myocardial infarction, transient ischemic attacks/stroke, clinically significant arrhythmia, congestive heart failure, or cardiac valve abnormalities;
* Type 1 diabetes mellitus;
* Insulin treated type 2 diabetes mellitus.
* Renal insufficiency.
* Liver insufficiency.
* Malignant disease within 5 years of screening;
* Has hypertension (sitting blood pressure > 140/90 mmHg at screening)
* History of rectal surgery.
* History of HIV, hepatitis B, hepatitis.
* Has used, in the last four weeks, drugs that may affect blood coagulation, such as Aspirin (at a dose above 250 mg/day), Warfarin, Sintrom, Enoxaparin, Nadroparin, Heparin, Clopidogrel, Ticlopidine.
* Use of tricyclic or monoamine-oxidase inhibors.
* Has upon physical examination a rectal deformation or signs of rectal disease such as fissure, bleeding hemorrhoids, fistula, infection or space occupying lesion.
* Unable to understand the use instruction for the coated suppository, as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
fecal incontinence | 2 weeks

SECONDARY OUTCOMES:
quality of life | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroeneterology dept, Asaf harofe Medical center, Zrifin, Israel